CLINICAL TRIAL: NCT07247214
Title: Investigation of Parameters Related to Pain Catastrophizing, Fear of Movement, Neck Awareness and Upper Extremity Functionality in Individuals With Chronic Neck Pain - a Cross-sectional Study
Brief Title: Pain, Fear of Movement, Neck Awareness and Upper Extremity Functionality in Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Assistant Professor, Hasan Kalyoncu University
Other Study IDs: 2025/095
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Neck Pain
Keywords: Chronic neck Pain; pain catastrophizing; kinesiophobia; neck awareness; functionality
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic neck pain group: Questionnaires to assess pain catastrophizing, kinesiophobia, neck awareness, and upper extremity functionality were administered to individuals with chronic neck pain.

SUMMARY:
Our study aims to investigate the parameters related to pain catastrophizing, fear of movement, neck awareness and upper extremity functionality in individuals with chronic neck pain - a cross-sectional study.

DETAILED DESCRIPTION:
Chronic neck pain (CNP) is a common musculoskeletal problem that persists for more than three months and negatively affects an individual's daily activities. Neck pain is a complex condition that occurs through the interaction of many factors. Age, gender, history of neck pain, other musculoskeletal problems, postural weakness, the presence of repetitive trauma, and the individual's social and psychosocial status can all influence the onset and course of neck pain. In addition, chronic neck pain causes impairments in body awareness, affecting the perception of the cervical region, and this triggers the development of fear of movement (kinesiophobia). Kinesiophobia causes the individual to avoid movement due to pain and can also lead to a decrease in upper extremity functionality. While studies examining these variables separately are common in the literature, to our knowledge, there is no study that includes these parameters together. In this context, our study; It aims to investigate the parameters related to pain catastrophizing, fear of movement, neck awareness and upper extremity functionality in individuals with chronic neck pain - a cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have had neck pain for 3 months or longer
* Those with no neurological findings
* Those who agree to participate in the study

Exclusion Criteria:

* Individuals with a history of fractures
* Those who have had cervical surgery
* Individuals who provide incomplete data
* Individuals who are inadequately literate in Turkish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who met the inclusion criteria and volunteered to participate in the study were administered the relevant assessment scales, which took approximately 30 minutes. No harmful practices or questions were posed to any participants during the study.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2025-07-20 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Pain Catastrophizing | through study completion, an average of 3 months
  The Pain Catastrophizing Scale (PCAT) will be used to assess pain catastrophizing. The PCAT, whose Turkish reliability and validity were established by Uğurlu et al., includes 13 situations describing different feelings and thoughts related to pain. Each situation is scored from 0 (never) to 4 (always). The total score ranges from 0 to 52 points. A higher total score indicates increased pain catastrophizing. According to the scale, individuals scoring 30 or higher are considered to have pain catastrophizing
Kinesiophobia | through study completion, an average of 3 months
  The Tampa Kinesiophobia Scale was used to assess fear of movement. The questionnaire, which will be used to measure individuals' perspectives on movement and their fear aspects, consists of 17 questions with total scores ranging from 17 to 68. Tampa scores greater than 37 indicate significant kinesiophobia.
Neck awareness | through study completion, an average of 3 months
  The Fremantle Neck Awareness Questionnaire was used to assess neck awareness. It is a simple Likert-type questionnaire (0 = I never feel like this, 1 = I rarely feel like this, 2 = I sometimes or some of the time feel like this, 3 = I often feel like this, 4 = I always or most of the time feel like this) that assesses individual perception. The questionnaire asks nine questions, including how individuals perceive their neck relative to their body and how they perceive their body position. A high score indicates poor awareness.
Upper extremity function | through study completion, an average of 3 months
  The Quick Questionnaire for Disabilities of the Arm, Shoulder, and Hand (Q-DASH) was used to assess individuals' upper extremity function. This 30-question questionnaire assesses an individual's ability to perform functional activities (21 items), pain (5 items), and psychosocial aspects of the disease (4 items). The total score ranges from 0 to 100, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
The pain | through study completion, an average of 3 months
  The short form of the McGill Pain Questionnaire (SF-MPQ) was used to assess pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 emotional) rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate, or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words selected for the sensory, emotional, and total descriptors. A higher score indicates a higher level of pain.
The pain | through study completion, an average of 3 months
  The Northwick Park Neck Pain Questionnaire was assessed. The Northwick Park Neck Pain Questionnaire is a multidimensional questionnaire consisting of nine items: neck pain intensity, sleep disturbance, numbness, duration of symptoms, and impairment in activities such as carrying heavy objects, reading and watching television, working, socializing, and driving. The driving item is optional. Each item has one question and five statements indicating increasing difficulty or pain. Responses to each question are scored from 0 to 4, with 4 representing the greatest impairment, and a total score is obtained by summing the scores for each of the nine items (possible scores: 0-36).

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba GÖNEN, Asisst. Prof. Dr., Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Candeniz S, Citaker S, Bakirarar B. Cross-cultural adaptation, reliability, and validity of the Turkish version of the Neck OutcOme Score. Turk J Med Sci. 2019 Dec 16;49(6):1707-1714. doi: 10.3906/sag-1907-87. PMID 31655517
- [Result] Yakut Y, Yakut E, Bayar K, Uygur F. Reliability and validity of the Turkish version short-form McGill pain questionnaire in patients with rheumatoid arthritis. Clin Rheumatol. 2007 Jul;26(7):1083-7. doi: 10.1007/s10067-006-0452-6. Epub 2006 Nov 15. PMID 17106618
- [Result] Lundwall A, Ryman A, Bjarnegard Sellius A, Mannerkorpi K. Pain requires processing - How the experience of pain is influenced by Basic Body Awareness Therapy in patients with long-term pain. J Bodyw Mov Ther. 2019 Oct;23(4):701-707. doi: 10.1016/j.jbmt.2019.02.006. Epub 2019 Feb 5. PMID 31733750
- [Result] Carroll LJ, Hogg-Johnson S, van der Velde G, Haldeman S, Holm LW, Carragee EJ, Hurwitz EL, Cote P, Nordin M, Peloso PM, Guzman J, Cassidy JD. Course and prognostic factors for neck pain in the general population: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S87-96. doi: 10.1016/j.jmpt.2008.11.013. PMID 19251079
- [Result] Haller H, Lauche R, Cramer H, Rampp T, Saha FJ, Ostermann T, Dobos G. Craniosacral Therapy for the Treatment of Chronic Neck Pain: A Randomized Sham-controlled Trial. Clin J Pain. 2016 May;32(5):441-9. doi: 10.1097/AJP.0000000000000290. PMID 26340656